CLINICAL TRIAL: NCT05234632
Title: A Prospective Study to Evaluate the Safety and Performance of PICO 14 in the Management of Acute and Chronic Wounds
Brief Title: Study to Evaluate the PICO 14 Negative Pressure Wound Therapy System in the Management of Acute and Chronic Wounds
Acronym: PICO14
Status: Terminated | Type: Observational
Why Stopped: Due to enrolment issues with dehisced and DFU's wounds
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PICO14.WND.PRO.2019.03
Record Dates: First submitted 2021-05-28; First posted 2022-02-10 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2023-12

CONDITIONS: Surgical Incision; Ulcer Foot; Ulcer Venous; Ulcer, Leg; Pressure Ulcer; Wound Dehiscence
Keywords: Closed incision wounds; Chronic wounds; PICO
MeSH Terms: conditions — Surgical Wound; Foot Ulcer; Varicose Ulcer; Leg Ulcer; Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PICO 14 Closed Incisions: Any Closed incision treated with PICO 14, for closed Surgical incisions this will be for 14 days post-surgery and with a 30 day follow up.
  Interventions: Device: PICO 14 single-use Negative Pressure Wound Therapy System
- PICO 14 Chronic/Dehisced Surgical Wounds: Any Chronic/Dehisced Surgical wound treated with PICO 14, for chronic and dehisced wounds this will be for up to 28 days therapy and no follow-up.
  Interventions: Device: PICO 14 single-use Negative Pressure Wound Therapy System

INTERVENTIONS:
Device: PICO 14 single-use Negative Pressure Wound Therapy System — The PICO14 device delivers negative pressure across the wound bed or closed incision and surrounding area, and exudate is managed by the dressing through a combination of absorption and evaporation of moisture through the outer film.

SUMMARY:
This is a prospective, multi-center, open label study evaluating the performance of PICO14 Negative Pressure Wound Therapy (NPWT) in the management of chronic open wounds (pressure ulcers, venous leg ulcers, diabetes related foot ulcers), dehisced surgical wounds and closed surgical incisions. The study comprises the Post Market Clinical Follow-up (PMCF) for a new variant of an established product. PICO 14 is based on another dressing called PICO.

The primary objective is to evaluate functional performance of PICO 14 through verification of delivery of negative pressure and wound exudate management.

ELIGIBILITY:
Inclusion Criteria:

* The subject must provide written informed consent.
* Subjects eighteen (18) years of age or older.
* Willing and able to make all required study visits.
* Able to follow instructions.
* Subject is suitable to participate in the study in the opinion of the Investigator.

Closed Incisions ONLY:

* Subject has a suitable, closed surgical incision which the clinician considers is suitable for PICO therapy, where it is expected that the therapy will be applied for up to 14 days.
* Any closed surgical incision in a patient in which the patient is deemed high risk of developing surgical site infection (SSI) in the opinion of the investigator.

Chronic wounds ONLY:

* Patients with any chronic wound* which the treating clinician deems is suitable for management with single-use disposable NPWT where it is expected that the therapy will applied for up to 28 days.

  * *Chronic wound in this study is defined as any wound of less than three months duration that is not healing after 4 weeks of standard care and having addressed the underlying cause.

Dehisced surgical wounds ONLY:

* Patients with dehisced wounds in which the clinician believes is suitable for PICO therapy where therapy is expected to be applied for up to 28 days.

  * *Wound dehiscence is a surgical complication in which two sides of a surgical incision separate and rupture along the incision, dehiscence typically is diagnosed after 2-3 days postsurgery and up to a month with more complicated surgeries

Exclusion Criteria:

* Contraindications (per the PICO 14 Instructions for use [IFU]) or hypersensitivity to the use of the investigational product or their components (e.g. silicone adhesives and polyurethane films [direct contact with incision], acrylic adhesives [direct contact with skin], polyethylene fabrics and super-absorbent powders [polyacrylates]) within the dressing).
* Subjects who require the use of SECURA non-sting barrier skin wipes and have hypersensitivity to the ingredients in the wipes.
* Participation in the treatment period of another clinical trial within thirty (30) days of operative visit or during the study.
* Subjects with skin features (e.g. tattoos, skin colour, preexisting scarring) which in the opinion of the Investigator, will interfere with the study assessments.
* Patients undergoing a procedure as part of palliative care (to be confirmed during surgery).
* Subjects who have participated previously in this clinical trial
* Subjects with a history of poor compliance with medical treatment.
* Malignant wounds, open abdomen, wounds which have been previously managed with NPWT in the previous four weeks.
* Pregnancy.
* Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.
* Presence of infection as determined by the clinical signs and symptoms (International wound infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seventy patients with Chronic open wounds (pressure ulcers, venous leg ulcers, diabetes-related foot ulcers, dehisced surgical wounds) and Closed surgical incisions, will be recruited to the study and will receive therapy with PICO 14. There will be a minimum of 10 of each of the following wound type; venous leg ulcers, diabetes-related foot ulcers, pressure ulcers, dehisced surgical wounds and post-operative incisions. The patients will be recruited from up to 7 sites in the United Kingdom, EU, and US, Canada. Sites failing to enroll may be replaced.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jahnke, Study Director — Smith & Nephew, Inc.
Locations (6):
- Klinikum der Landeshauptstadt Stuttgart gKAöR, Stuttgart, Germany
- United Kingdom (5):
  - Queen Elizabeth the Queen Mother Hospital, Margate
  - Northumbria Healthcare NHS Trust, Newcastle
  - Nottingham Breast Institute, Nottingham
  - Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry
  - The Lantern Centre, Preston

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 45 participants were enrolled to the study at 6 sites. There was one (1) screen failure, leaving 44 subjects (25 closed incisions; 19 chronic wounds) receiving PICO 14 NPWT treatment forming the safety analysis set (SAF).
Period: Overall Study
Arm/Group | PICO 14 Closed Incisions | PICO 14 Chronic/Dehisced Surgical Wounds
Started | 25 | 19
Completed | 20 | 13
Not Completed | 5 | 6
Not completed — Participant Withdrawn: Non-Compliance | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 0 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Participant tested positive for COVID-19 and is in isolation | 0 | 1
Not completed — Withdrawn by participant upon experiencing Adverse Event. | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received the study device with available data.
Groups:
- Total: Total of all reporting groups
Arm/Group | PICO 14 Closed Incisions | PICO 14 Chronic/Dehisced Surgical Wounds | Total
Number analyzed (Participants) | 25 | 19 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (10.2) | 71.3 (16.3) | 71.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 25 | 15 | 40
  Race: Black | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0
  Race: Other | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25 | 16 | 41
  Germany | 0 | 3 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (4.6) | 30.0 (9.8) | 29.5 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Delivery of Nominal -80mmHg Negative Pressure
Description: Delivery of nominal -80mmHg negative pressure over the treatment period was measured by download of the built-in data chip from the PICO 14 devices to collect NPWT delivery status. This data was summarized to provide the average negative pressure delivery overall and for both closed incisions and chronic/dehisced surgical wounds.
Time Frame: Day 30
Population: Full Analysis Set (FAS) population included all participants recruited into the study that attended at least one post-baseline assessment with available data at the time frame indicated.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Groups:
- PICO 14 Overall (Closed Incisions & Chronic/Dehisced Wounds): Any wound treated with PICO 14. For closed Surgical incisions this will be for 14 days post surgery and with a 30 day follow up. For chronic and dehisced wounds this will be for up to 28 days therapy and no follow-up.
  PICO 14 single-use Negative Pressure Wound Therapy System: The PICO14 device delivers negative pressure across the wound bed or closed incision and surrounding area, and exudate is managed by the dressing through a combination of absorption and evaporation of moisture through the outer film.
Arm/Group | PICO 14 Closed Incisions | PICO 14 Chronic/Dehisced Surgical Wounds | PICO 14 Overall (Closed Incisions & Chronic/Dehisced Wounds)
Number analyzed (Participants) | 18 | 13 | 31
millimeters of mercury (mmHg) | -77.2 (7.7) | -74.7 (11.4) | -76.2 (9.3)

2. Primary Outcome: Exudate Management: Occurrence of No Exudate Leaks
Description: Exudate management was measured by the number of participants with no exudate leaks identified by the clinician at any point over the treatment period, up to 30 days.
Time Frame: Up to 30 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Closed Incisions | PICO 14 Chronic/Dehisced Surgical Wounds | PICO 14 Overall (Closed Incisions & Chronic/Dehisced Wounds)
Number analyzed (Participants) | 20 | 13 | 33
Participants | 13 | 8 | 21

3. Secondary Outcome: Scar Quality Measured by The Patient and Observer Scar Assessment Scale (POSAS): Closed Incision Only
Description: The Patient and Observer Scar Assessment Scale (POSAS) is a comprehensive scale that is designed for the evaluation of all types of scars by professionals and patients. The POSAS consists of two parts: a Patient Scale and an Observer Scale. Both scales contain six items that are scored numerically and make up a 'Total Score' of the Patient and Observer Scale.
  Each item of both scales has a 10-point score, with 10 indicating the worst imaginable scar or sensation. The lowest score is '1', and corresponds to the situation of normal skin (normal pigmentation, no itching etc.), and goes up to the worst imaginable. The Total Score is provided for both the Patient Scale and Observer Scale at Day 14 & Day 30. The Total Score for both scales was calculated by summing up the scores of each of the six items. The Total Score ranged from 6 to 60 with a lower score indicating a better outcome.
Time Frame: Day 14 and Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 20
score on a scale
  Day 14: Patient Scale Total Score: number analyzed (Participants) | 18
  Day 14: Patient Scale Total Score | 18.9 (11.9)
  Day 14: Observer Scale Total Score: number analyzed (Participants) | 19
  Day 14: Observer Scale Total Score | 16.3 (9)
  Day 30: Patient Scale Total Score | 19.5 (10.6)
  Day 30: Observer Scale Total Score: number analyzed (Participants) | 19
  Day 30: Observer Scale Total Score | 13.7 (7.4)

4. Secondary Outcome: Number of Participants With Surgical Site Infections (SSC): Closed Incisions Only
Description: Incidence of Surgical Site Infections (SSI) as defined by The Centers for Disease Control and Prevention (CDC) criteria, for any incision that had not healed by the given assessment at Day 7, Day 14, and Day 30. The number of participants with an incision that is clinically infected were categorized as either 'Yes' or 'No' (e.g., Is Incision Clinically Infected: Yes or No).
Time Frame: Day 7, Day 14, and Day 30
Population: Full Analysis Set (FAS) population included all participants recruited into the study that attended at least one post-baseline assessment with available data at the time frame indicated.
  The FAS population for this outcome measure includes only participants with Closed Incisions identified as not healed (i.e., not fully closed/epithelialized).
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 8
Participants
  Day 7: Is Incision Clinically Infected: Yes | 0
  Day 7: Is Incision Clinically Infected: No | 8
  Day 14: Is Incision Clinically Infected: number analyzed (Participants) | 2
  Day 14: Is Incision Clinically Infected: Yes | 2
  Day 14: Is Incision Clinically Infected: No | 0
  Day 30: Is Incision Clinically Infected: number analyzed (Participants) | 2
  Day 30: Is Incision Clinically Infected: Yes | 0
  Day 30: Is Incision Clinically Infected: No | 2

5. Secondary Outcome: Number of Participants With Surgical Site Complication (SSC): Closed Incisions Only
Description: Incidence of Surgical Site Complication (SSC) for any incision that had not healed by the given assessment at Day 7, Day 14, and Day 30. The number of participants where dehiscence of incision occurred, were categorized as either 'Yes' or 'No' (e.g., Incision dehisced: Yes or No).
Time Frame: Day 7, Day 14, and Day 30
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 8
Participants
  Day 7: Incision Dehisced: Yes | 0
  Day 7: Incision Dehisced: No | 8
  Day 14: Incision Dehisced: number analyzed (Participants) | 2
  Day 14: Incision Dehisced: Yes | 1
  Day 14: Incision Dehisced: No | 1
  Day 30: Incision Dehisced: number analyzed (Participants) | 2
  Day 30: Incision Dehisced: Yes | 1
  Day 30: Incision Dehisced: No | 1

6. Secondary Outcome: Condition of Peri-Wound Skin Assessed Through Visual Inspection at 7, 14 and 30 Days: Closed Incisions Only
Description: The clinician assessed the condition of the surrounding skin of closed incisions at Day 7, Day 14, and Day 30. The condition of skin was categorized as the number of participants where any of the following characteristics apply:
  * Healthy
  * Fragile
  * Inflamed
  * Erythematous
  * Oedematous
  * Eczematous
  * Macerated
  * Bruising
  * Dry and flaky
  * Other
Time Frame: Day 7, Day 14, and Day 30
Population: Full Analysis Set (FAS) population included all participants recruited into the study that attended at least one post-baseline assessment with available data at the time frame indicated for Closed Incisions only.
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 22
Participants
  Day 7: Healthy | 18
  Day 7: Fragile | 0
  Day 7: Inflamed | 0
  Day 7: Erythematous | 0
  Day 7: Oedematous | 0
  Day 7: Eczematous | 0
  Day 7: Macerated | 0
  Day 7: Bruising | 11
  Day 7: Dry and flaky | 0
  Day 7: Other | 0
  Day 14: Healthy: number analyzed (Participants) | 20
  Day 14: Healthy | 15
  Day 14: Fragile: number analyzed (Participants) | 20
  Day 14: Fragile | 1
  Day 14: Inflamed: number analyzed (Participants) | 20
  Day 14: Inflamed | 1
  Day 14: Erythematous: number analyzed (Participants) | 20
  Day 14: Erythematous | 2
  Day 14: Oedematous: number analyzed (Participants) | 20
  Day 14: Oedematous | 1
  Day 14: Eczematous: number analyzed (Participants) | 20
  Day 14: Eczematous | 0
  Day 14: Macerated: number analyzed (Participants) | 20
  Day 14: Macerated | 2
  Day 14: Bruising: number analyzed (Participants) | 20
  Day 14: Bruising | 4
  Day 14: Dry and flaky: number analyzed (Participants) | 20
  Day 14: Dry and flaky | 1
  Day 14: Other: number analyzed (Participants) | 20
  Day 14: Other | 0
  Day 30: Healthy: number analyzed (Participants) | 20
  Day 30: Healthy | 20
  Day 30: Fragile: number analyzed (Participants) | 20
  Day 30: Fragile | 0
  Day 30: Inflamed: number analyzed (Participants) | 20
  Day 30: Inflamed | 0
  Day 30: Erythematous: number analyzed (Participants) | 20
  Day 30: Erythematous | 1
  Day 30: Oedematous: number analyzed (Participants) | 20
  Day 30: Oedematous | 0
  Day 30: Eczematous: number analyzed (Participants) | 20
  Day 30: Eczematous | 0
  Day 30: Macerated: number analyzed (Participants) | 20
  Day 30: Macerated | 1
  Day 30: Bruising: number analyzed (Participants) | 20
  Day 30: Bruising | 0
  Day 30: Dry and flaky: number analyzed (Participants) | 20
  Day 30: Dry and flaky | 1
  Day 30: Other: number analyzed (Participants) | 20
  Day 30: Other | 0

7. Secondary Outcome: Level of Pain - Visual Analog Score (VAS): Closed Incisions Only
Description: Level of pain on dressing application, during wear and at dressing removal assessed by Visual Analog Score (VAS) scale over the 14 day treatment period. The VAS scale ranges from 0-10 with 0 being no pain and 10 being extreme pain.
Time Frame: Up to 14 Days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Dressings
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 22
Number analyzed (Dressings) | 47
score on a scale
  Level of Pain: Dressing Application: number analyzed (Dressings) | 26
  Level of Pain: Dressing Application | 0.5 (1.3)
  Level of Pain: During Wear: number analyzed (Dressings) | 46
  Level of Pain: During Wear | 2.5 (2.5)
  Level of Pain: Dressing Removal | 1.3 (1.9)

8. Secondary Outcome: Patient Satisfaction During Wear - Performance: Closed Incisions Only
Description: Patient satisfaction in performance at Day 7, Day 14, and Day 30 (follow-up) measured by response of 'Yes' or 'No' to the following:
  * Overall performance
  * Comfort during wear
  * Noise level
  * Discreetness
  * Portability
Time Frame: Day 7, Day 14, and Day 30
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 20
Participants
  Day 7: Overall performance: Yes | 20
  Day 7: Overall performance: No | 0
  Day 7: Comfort during wear: Yes | 19
  Day 7: Comfort during wear: No | 1
  Day 7: Noise level: Yes | 18
  Day 7: Noise level: No | 2
  Day 7: Discreetness: Yes | 20
  Day 7: Discreetness: No | 0
  Day 7: Portability: Yes | 18
  Day 7: Portability: No | 2
  Day 14: Overall performance: number analyzed (Participants) | 19
  Day 14: Overall performance: Yes | 18
  Day 14: Overall performance: No | 1
  Day 14: Comfort during wear: number analyzed (Participants) | 19
  Day 14: Comfort during wear: Yes | 16
  Day 14: Comfort during wear: No | 3
  Day 14: Noise level: number analyzed (Participants) | 19
  Day 14: Noise level: Yes | 16
  Day 14: Noise level: No | 3
  Day 14: Discreetness: number analyzed (Participants) | 19
  Day 14: Discreetness: Yes | 17
  Day 14: Discreetness: No | 2
  Day 14: Portability: number analyzed (Participants) | 19
  Day 14: Portability: Yes | 13
  Day 14: Portability: No | 6
  Day 30: Overall performance: number analyzed (Participants) | 13
  Day 30: Overall performance: Yes | 13
  Day 30: Overall performance: No | 0
  Day 30: Comfort during wear: number analyzed (Participants) | 13
  Day 30: Comfort during wear: Yes | 11
  Day 30: Comfort during wear: No | 2
  Day 30: Noise level: number analyzed (Participants) | 13
  Day 30: Noise level: Yes | 10
  Day 30: Noise level: No | 3
  Day 30: Discreetness: number analyzed (Participants) | 13
  Day 30: Discreetness: Yes | 13
  Day 30: Discreetness: No | 0
  Day 30: Portability: number analyzed (Participants) | 13
  Day 30: Portability: Yes | 12
  Day 30: Portability: No | 1

9. Secondary Outcome: Patient Satisfaction During Wear - Interference With Daily Living: Closed Incisions Only
Description: Patient satisfaction during wear in interference with daily living at Day 7, Day 14, and Day 30 (follow-up) measured by response of 'Yes' or 'No' to the following:
  * Showering
  * Sleeping
  * Socializing
  * Working
Time Frame: Day 7, Day 14, and Day 30
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 20
Participants
  Day 7: Showering: number analyzed (Participants) | 11
  Day 7: Showering: Yes | 8
  Day 7: Showering: No | 3
  Day 7: Sleeping: Yes | 18
  Day 7: Sleeping: No | 2
  Day 7: Socializing: number analyzed (Participants) | 13
  Day 7: Socializing: Yes | 13
  Day 7: Socializing: No | 0
  Day 7: Working: number analyzed (Participants) | 3
  Day 7: Working: Yes | 2
  Day 7: Working: No | 1
  Day 14: Showering: number analyzed (Participants) | 13
  Day 14: Showering: Yes | 10
  Day 14: Showering: No | 3
  Day 14: Sleeping: number analyzed (Participants) | 19
  Day 14: Sleeping: Yes | 16
  Day 14: Sleeping: No | 3
  Day 14: Socializing: number analyzed (Participants) | 16
  Day 14: Socializing: Yes | 16
  Day 14: Socializing: No | 0
  Day 14: Working: number analyzed (Participants) | 5
  Day 14: Working: Yes | 2
  Day 14: Working: No | 3
  Day 30: Showering: number analyzed (Participants) | 7
  Day 30: Showering: Yes | 5
  Day 30: Showering: No | 2
  Day 30: Sleeping: number analyzed (Participants) | 13
  Day 30: Sleeping: Yes | 11
  Day 30: Sleeping: No | 2
  Day 30: Socializing: number analyzed (Participants) | 12
  Day 30: Socializing: Yes | 11
  Day 30: Socializing: No | 1
  Day 30: Working: number analyzed (Participants) | 5
  Day 30: Working: Yes | 4
  Day 30: Working: No | 1

10. Secondary Outcome: Ease of Application and Removal: Closed Incisions Only
Description: Ease of application and removal of the PICO 14 dressing for Closed Incisions determined by overall count of dressings applied/removed based on responses to the questions "Was it easy to apply the dressing" and "Was it easy to remove the dressing" as either 'Yes' or 'No'.
Time Frame: Up to 14 days
Population: as for outcome 6
Measure: Count of Units; unit: dressings
Units Other Than Participants: dressings
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 22
Number analyzed (dressings) | 48
dressings
  Was it easy to apply the dressing: Yes | 48
  Was it easy to apply the dressing: No | 0
  Was it easy to remove the dressing: Yes | 46
  Was it easy to remove the dressing: No | 2

11. Secondary Outcome: Dressing Wear Time: Closed Incisions Only
Description: Overall dressing wear time in days for Closed Incisions only.
Time Frame: Up to 14 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: dressings
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 22
Number analyzed (dressings) | 51
days | 5.7 (2.1)

12. Secondary Outcome: Dressing Conformability: Closed Incisions Only
Description: Dressing conformability to the closed incision wound measured by the number of responses to the question "Was the dressing conformable on the incision/wound?" as either 'Yes' or 'No'.
Time Frame: Up to 14 days
Population: as for outcome 6
Measure: Count of Units; unit: dressings
Units Other Than Participants: dressings
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 22
Number analyzed (dressings) | 48
dressings
  Yes | 48
  No | 0

13. Secondary Outcome: Number of Dressings Used: Closed Incisions Only
Description: Dressing change frequency summarized as the number of dressings used per participants for Closed Incisions.
Time Frame: Up to 14 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: dressings per participant
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 22
dressings per participant | 2.2 (1.0)

14. Secondary Outcome: Reason for Dressing Change: Closed Incisions Only
Description: Reason for dressing change for Closed Incisions only. Count of occurrences by dressing were categorized as 'Yes' or 'No':
  * Routine dressing change
  * Inadequate exudate management
  * Pain/discomfort
  * Dressing damaged
  * Dressing fell off
  * Patient removed dressing
  * Adverse Event
  * Surgical procedure
  * Safety alarm
  * Dressing components not in place
  * No vacuum
  * other
Time Frame: Up to 14 days
Population: as for outcome 6
Measure: Count of Units; unit: dressings
Units Other Than Participants: dressings
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 22
Number analyzed (dressings) | 51
dressings
  Routine dressing change: Yes | 37
  Routine dressing change: No | 14
  Inadequate exudate management: Yes | 5
  Inadequate exudate management: No | 46
  Pain/discomfort: Yes | 0
  Pain/discomfort: No | 51
  Dressing damaged: Yes | 0
  Dressing damaged: No | 51
  Dressing fell off: Yes | 0
  Dressing fell off: No | 51
  Patient removed dressing: Yes | 1
  Patient removed dressing: No | 50
  Adverse Event: Yes | 4
  Adverse Event: No | 47
  Surgical procedure: Yes | 0
  Surgical procedure: No | 51
  Safety alarm: Yes | 1
  Safety alarm: No | 50
  Dressing components not in place: Yes | 1
  Dressing components not in place: No | 50
  No vacuum: Yes | 2
  No vacuum: No | 49
  Other: Yes | 3
  Other: No | 48

15. Secondary Outcome: Clinician Acceptability of PICO 14 at Discontinuation of Therapy: Closed Incision Only
Description: Acceptability of the device determined from the clinician's response (Yes/No) at discontinuation of therapy by participant (i.e., Day 14) to the question: Overall are you satisfied with the performance of the PICO 14 system (pump and PICO 14 dressing)?
Time Frame: Day 14
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Closed Incisions
Number analyzed (Participants) | 19
Participants
  Yes | 19
  No | 0

16. Secondary Outcome: Number of Participants With Clinical Infection: Chronic and Dehisced Surgical Wounds Only
Description: Count of participants with presence of infection as determined by the clinical signs and symptoms at Day 0, Day 7, Day 14, Day 21, and Day 28 for Chronic and Dehisced Surgical Wounds (i.e., clinically infected: 'Yes' or 'No').
Time Frame: Day 0, Day 7, Day 14, Day 21, and Day 28
Population: Full Analysis Set (FAS) population included all participants recruited into the study that attended at least one post-baseline assessment with available data at the time frame indicated for Chronic and Dehisced Surgical Wounds only.
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Participants
  Day 0: Clinically infected: Yes | 0
  Day 0: Clinically infected: No | 16
  Day 7: Clinically infected: Yes | 0
  Day 7: Clinically infected: No | 16
  Day 14: Clinically infected: number analyzed (Participants) | 15
  Day 14: Clinically infected: Yes | 0
  Day 14: Clinically infected: No | 15
  Day 21: Clinically infected: number analyzed (Participants) | 14
  Day 21: Clinically infected: Yes | 0
  Day 21: Clinically infected: No | 14
  Day 28: Clinically infected: number analyzed (Participants) | 13
  Day 28: Clinically infected: Yes | 0
  Day 28: Clinically infected: No | 13

17. Secondary Outcome: Appearance of the Wound by Size: Chronic and Dehisced Surgical Wounds Only
Description: Appearance of the wound by size measured by the length and width in centimeters at screening and Day 28 for Chronic and Dehisced Surgical Wounds only.
Time Frame: Screening and Day 28
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
centimeters (cm)
  Screening: Length | 5.9 (5.2)
  Day 28: Length: number analyzed (Participants) | 13
  Day 28: Length | 3.1 (2.2)
  Screening: Width | 4.5 (2.9)
  Day 28: Width: number analyzed (Participants) | 13
  Day 28: Width | 3.1 (2.4)

18. Secondary Outcome: Appearance of the Wound by Depth: Chronic and Dehisced Surgical Wounds Only
Description: Appearance of the wound by depth measured in millimeters at screening and Day 28 for Chronic and Dehisced Surgical Wounds only.
Time Frame: Screening and Day 28
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
millimeters (mm)
  Screening: Depth | 10.6 (11.1)
  Day 28: Depth: number analyzed (Participants) | 12
  Day 28: Depth | 3.2 (5.7)

19. Secondary Outcome: Appearance of the Wound by Presence of Necrotic Tissue: Chronic and Dehisced Surgical Wounds Only
Description: Appearance of the wound by number of participants with the presence of necrotic tissue (Yes/No) at screening and Day 28 for Chronic and Dehisced Surgical Wounds.
Time Frame: Screening and Day 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Participants
  Screening: Presence of Necrotic Tissue: Yes | 8
  Screening: Presence of Necrotic Tissue: No | 8
  Day 28: Presence of Necrotic Tissue: number analyzed (Participants) | 13
  Day 28: Presence of Necrotic Tissue: Yes | 3
  Day 28: Presence of Necrotic Tissue: No | 10

20. Secondary Outcome: Appearance of the Wound by Necrotic Tissue Amount: Chronic and Dehisced Surgical Wounds Only
Description: Appearance of the wound by amount of necrotic tissue at screening and Day 28 for Chronic and Dehisced Surgical Wounds categorized as number of participants with:
  * <25% of wound bed covered
  * 25% to 50% of wound covered
  * 50% to < 75% of wound covered
  * 75% to 100% of wound covered
Time Frame: Screening and Day 28
Population: Full Analysis Set (FAS) population included all participants recruited into the study that attended at least one post-baseline assessment with available data at the time frame indicated for Chronic and Dehisced Surgical Wounds with presence of necrotic tissue only.
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 8
Participants
  Screening: Necrotic Tissue Amount: <25% of wound bed covered | 5
  Screening: Necrotic Tissue Amount: 25% to 50% of wound covered | 2
  Screening: Necrotic Tissue Amount: 50% to < 75% of wound covered | 1
  Screening: Necrotic Tissue Amount: 75% to 100% of wound covered | 0
  Day 28: Necrotic Tissue Amount: number analyzed (Participants) | 3
  Day 28: Necrotic Tissue Amount: <25% of wound bed covered | 2
  Day 28: Necrotic Tissue Amount: 25% to 50% of wound covered | 0
  Day 28: Necrotic Tissue Amount: 50% to < 75% of wound covered | 1
  Day 28: Necrotic Tissue Amount: 75% to 100% of wound covered | 0

21. Secondary Outcome: Appearance of the Wound by Type of Necrotic Tissue: Chronic and Dehisced Surgical Wounds Only
Description: Appearance of the wound by type of necrotic tissue at screening and Day 28 for Chronic and Dehisced Surgical Wounds categorized as number of participants with:
  * White/grey non-viable tissue
  * Non-adherent, yellow slough
  * Loosely adherent, yellow slough
  * Adherent, soft, black eschar
  * Firmly adherent, hard/black eschar
Time Frame: Screening and Day 28
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 8
Participants
  Screening: Type of Necrotic Tissue: White/grey non-viable tissue | 0
  Screening: Type of Necrotic Tissue: Non-adherent, yellow slough | 3
  Screening: Type of Necrotic Tissue: Loosely adherent, yellow slough | 5
  Screening: Type of Necrotic Tissue: Adherent, soft, black eschar | 0
  Screening: Type of Necrotic Tissue: Firmly adherent, hard/black eschar | 0
  Day 28: Type of Necrotic Tissue: number analyzed (Participants) | 3
  Day 28: Type of Necrotic Tissue: White/grey non-viable tissue | 0
  Day 28: Type of Necrotic Tissue: Non-adherent, yellow slough | 1
  Day 28: Type of Necrotic Tissue: Loosely adherent, yellow slough | 2
  Day 28: Type of Necrotic Tissue: Adherent, soft, black eschar | 0
  Day 28: Type of Necrotic Tissue: Firmly adherent, hard/black eschar | 0

22. Secondary Outcome: Appearance of the Wound by Granulation Tissue: Chronic and Dehisced Surgical Wounds Only
Description: Appearance of the wound by granulation tissue at screening and Day 28 for Chronic and Dehisced Surgical Wounds categorized as number of participants with:
  * Skin intact or partial thickness wound
  * Bright, beefy red; 75% to 100% of wound filled &/or tissue overgrowth
  * Bright, beefy red; < 75% & >25% of wound filled
  * Pink, &/or dull, dusky red &/or fills <25% of wound
  * No granulation tissue present
Time Frame: Screening and Day 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Participants
  Screening: Granulation Tissue: Skin intact or partial thickness wound | 0
  Screening: Granulation Tissue: Bright, beefy red; 75% to 100% of wound filled &/or tissue overgrowth | 7
  Screening: Granulation Tissue: Bright, beefy red; < 75% & >25% of wound filled | 6
  Screening: Granulation Tissue: Pink, &/or dull, dusky red &/or fills <25% of wound | 3
  Screening: Granulation Tissue: No granulation tissue present | 0
  Day 28: Granulation Tissue: number analyzed (Participants) | 13
  Day 28: Granulation Tissue: Skin intact or partial thickness wound | 1
  Day 28: Granulation Tissue: Bright, beefy red; 75% to 100% of wound filled &/or tissue overgrowth | 5
  Day 28: Granulation Tissue: Bright, beefy red; < 75% & >25% of wound filled | 6
  Day 28: Granulation Tissue: Pink, &/or dull, dusky red &/or fills <25% of wound | 1
  Day 28: Granulation Tissue: No granulation tissue present | 0

23. Secondary Outcome: Appearance of the Wound by Epithelialization: Chronic and Dehisced Surgical Wounds Only
Description: Appearance of the wound by epithelialization at screening and Day 28 for Chronic and Dehisced Surgical Wounds categorized as number of participants with:
  * 100% wound covered, surface intact
  * 75% to < 100% wound covered &/or epithelial tissue extends to > 0.5 cm into wound bed
  * 50% to < 75% wound covered &/or epithelial tissue extends to < 0.5 cm into wound bed
  * 25% to < 50% wound covered
  * < 25% wound covered
Time Frame: Screening and Day 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Participants
  Screening: Epithelialization: 100% wound covered, surface intact | 0
  Screening: Epithelialization: 75% to < 100% wound covered &/or epithelial tissue extends to > 0.5 cm into wound bed | 0
  Screening: Epithelialization: 50% to < 75% wound covered &/or epithelial tissue extends to < 0.5 cm into wound bed | 0
  Screening: Epithelialization: 25% to < 50% wound covered | 0
  Screening: Epithelialization: < 25% wound covered | 16
  Day 28: Epithelialization: number analyzed (Participants) | 13
  Day 28: Epithelialization: 100% wound covered, surface intact | 0
  Day 28: Epithelialization: 75% to < 100% wound covered &/or epithelial tissue extends to > 0.5 cm into wound bed | 1
  Day 28: Epithelialization: 50% to < 75% wound covered &/or epithelial tissue extends to < 0.5 cm into wound bed | 1
  Day 28: Epithelialization: 25% to < 50% wound covered | 2
  Day 28: Epithelialization: < 25% wound covered | 9

24. Secondary Outcome: Appearance of the Wound by Presence of Exudate: Chronic and Dehisced Surgical Wounds Only
Description: Appearance of the wound by number of participants with presence of exudate (Yes/No) at screening and Day 28 for Chronic and Dehisced Surgical Wounds.
Time Frame: Screening and Day 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Participants
  Screening: Presence of Exudate: Yes | 15
  Screening: Presence of Exudate: No | 1
  Day 28: Presence of Exudate: number analyzed (Participants) | 13
  Day 28: Presence of Exudate: Yes | 12
  Day 28: Presence of Exudate: No | 1

25. Secondary Outcome: Appearance of the Wound by Level of Exudate: Chronic and Dehisced Surgical Wounds Only
Description: Appearance of the wound by number of participants level of exudate at screening and Day 28 for Chronic and Dehisced Surgical Wounds categorized as:
  * Light
  * Moderate
  * Heavy
Time Frame: Screening and Day 28
Population: Full Analysis Set (FAS) population included all participants recruited into the study that attended at least one post-baseline assessment with available data at the time frame indicated for Chronic and Dehisced Surgical Wounds with exudate present only.
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 15
Participants
  Screening: Level of Exudate: Light | 2
  Screening: Level of Exudate: Moderate | 12
  Screening: Level of Exudate: Heavy | 1
  Day 28: Level of Exudate: number analyzed (Participants) | 12
  Day 28: Level of Exudate: Light | 6
  Day 28: Level of Exudate: Moderate | 5
  Day 28: Level of Exudate: Heavy | 1

26. Secondary Outcome: Condition of Peri-Wound Skin Assessed Through Visual Inspection at Day 0, Day 7, Day 14, Day 21, and Day 28 Days: Chronic and Dehisced Surgical Wounds Only
Description: The clinician assessed the condition of the surrounding skin of Chronic and Dehisced Surgical Wounds at Day 0, Day 7, Day 14, Day 21, and Day 28. The condition of skin was categorized as the number of participants where any of the following characteristics apply:
  * Normal
  * Erythematous
  * Oedematous
  * Eczematous
  * Excoriated
  * Macerated
  * Indurated
  * Other
Time Frame: Day 0, Day 7, Day 14, Day 21, and Day 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Participants
  Day 0 : Normal | 7
  Day 0 : Erythematous | 2
  Day 0 : Oedematous | 4
  Day 0 : Eczematous | 0
  Day 0 : Excoriated | 1
  Day 0 : Macerated | 3
  Day 0 : Indurated | 0
  Day 0 : Other | 2
  Day 7 : Normal | 6
  Day 7 : Erythematous | 2
  Day 7 : Oedematous | 3
  Day 7 : Eczematous | 0
  Day 7 : Excoriated | 1
  Day 7 : Macerated | 5
  Day 7 : Indurated | 0
  Day 7 : Other | 4
  Day 14 : Normal: number analyzed (Participants) | 15
  Day 14 : Normal | 5
  Day 14 : Erythematous: number analyzed (Participants) | 15
  Day 14 : Erythematous | 3
  Day 14 : Oedematous: number analyzed (Participants) | 15
  Day 14 : Oedematous | 3
  Day 14 : Eczematous: number analyzed (Participants) | 15
  Day 14 : Eczematous | 0
  Day 14 : Excoriated: number analyzed (Participants) | 15
  Day 14 : Excoriated | 3
  Day 14 : Macerated: number analyzed (Participants) | 15
  Day 14 : Macerated | 5
  Day 14 : Indurated: number analyzed (Participants) | 15
  Day 14 : Indurated | 0
  Day 14 : Other: number analyzed (Participants) | 15
  Day 14 : Other | 3
  Day 21 : Normal: number analyzed (Participants) | 14
  Day 21 : Normal | 5
  Day 21 : Erythematous: number analyzed (Participants) | 14
  Day 21 : Erythematous | 1
  Day 21 : Oedematous: number analyzed (Participants) | 14
  Day 21 : Oedematous | 2
  Day 21 : Eczematous: number analyzed (Participants) | 14
  Day 21 : Eczematous | 1
  Day 21 : Excoriated: number analyzed (Participants) | 14
  Day 21 : Excoriated | 1
  Day 21 : Macerated: number analyzed (Participants) | 14
  Day 21 : Macerated | 4
  Day 21 : Indurated: number analyzed (Participants) | 14
  Day 21 : Indurated | 0
  Day 21 : Other: number analyzed (Participants) | 14
  Day 21 : Other | 5
  Day 28 : Normal: number analyzed (Participants) | 13
  Day 28 : Normal | 4
  Day 28 : Erythematous: number analyzed (Participants) | 13
  Day 28 : Erythematous | 1
  Day 28 : Oedematous: number analyzed (Participants) | 13
  Day 28 : Oedematous | 1
  Day 28 : Eczematous: number analyzed (Participants) | 13
  Day 28 : Eczematous | 0
  Day 28 : Excoriated: number analyzed (Participants) | 13
  Day 28 : Excoriated | 2
  Day 28 : Macerated: number analyzed (Participants) | 13
  Day 28 : Macerated | 4
  Day 28 : Indurated: number analyzed (Participants) | 13
  Day 28 : Indurated | 0
  Day 28 : Other: number analyzed (Participants) | 13
  Day 28 : Other | 3

27. Secondary Outcome: Percentage Change in Area of Wound: Chronic and Dehisced Surgical Wounds Only
Description: The reference wound area captured at each study visit. Percentage change in area calculated and summarized using a Wilcoxon Signed Rank test from baseline to all post-baseline study visits at Day 7, Day 14, Day 21, and Day 28.
Time Frame: Day 7, Day 14, Day 21, and Day 28
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change in wound area
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
percent change in wound area
  Day 7 | 17.5 (24.7)
  Day 14: number analyzed (Participants) | 15
  Day 14 | 18.6 (31.0)
  Day 21: number analyzed (Participants) | 14
  Day 21 | 42.2 (22.7)
  Day 28: number analyzed (Participants) | 13
  Day 28 | 50.5 (24.0)

28. Secondary Outcome: Percentage Change in Volume of Wound: Chronic and Dehisced Surgical Wounds Only
Description: The reference wound volume captured at each study visit. Percentage change in volume calculated and summarized using a Wilcoxon Signed Rank test from baseline to all post-baseline study visits at Day 7, Day 14, Day 21, and Day 28.
Time Frame: Day 7, Day 14, Day 21, and Day 28
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change in wound volume
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 15
percent change in wound volume
  Day 7 | 41.8 (30.3)
  Day 14: number analyzed (Participants) | 14
  Day 14 | 52.3 (32.8)
  Day 21: number analyzed (Participants) | 13
  Day 21 | 72.7 (30.8)
  Day 28: number analyzed (Participants) | 11
  Day 28 | 79.3 (24.7)

29. Secondary Outcome: Level of Pain - Visual Analog Score (VAS): Chronic and Dehisced Surgical Wounds Only
Description: Level of pain on application, during wear and at dressing removal assessed by Visual Analog Score (VAS) scale over the 28 day treatment period. The VAS scale ranges from 0-10 with 0 being no pain and 10 being extreme pain.
Time Frame: Up to 28 days
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Number analyzed (dressings) | 99
score on a scale
  Level of Pain: Dressing Application: number analyzed (dressings) | 98
  Level of Pain: Dressing Application | 0.4 (1.4)
  Level of Pain: During Wear | 1.1 (2.1)
  Level of Pain: Dressing Removal: number analyzed (dressings) | 96
  Level of Pain: Dressing Removal | 1.5 (2.4)

30. Secondary Outcome: Patient Satisfaction During Wear - Performance: Chronic and Dehisced Surgical Wounds Only
Description: Patient satisfaction in performance at Day 14 and Day 28 measured by response of 'Yes' or 'No' to the following:
  * Overall performance
  * Comfort during wear
  * Noise level
  * Discreetness
  * Portability
Time Frame: Day 14 and Day 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 15
Participants
  Day 14: Overall performance: Yes | 15
  Day 14: Overall performance: No | 0
  Day 14: Comfort during wear: Yes | 15
  Day 14: Comfort during wear: No | 0
  Day 14: Noise level: Yes | 15
  Day 14: Noise level: No | 0
  Day 14: Discreetness: Yes | 15
  Day 14: Discreetness: No | 0
  Day 14: Portability: Yes | 15
  Day 14: Portability: No | 0
  Day 28: Overall performance: number analyzed (Participants) | 13
  Day 28: Overall performance: Yes | 13
  Day 28: Overall performance: No | 0
  Day 28: Comfort during wear: number analyzed (Participants) | 13
  Day 28: Comfort during wear: Yes | 13
  Day 28: Comfort during wear: No | 0
  Day 28: Noise level: number analyzed (Participants) | 13
  Day 28: Noise level: Yes | 13
  Day 28: Noise level: No | 0
  Day 28: Discreetness: number analyzed (Participants) | 13
  Day 28: Discreetness: Yes | 13
  Day 28: Discreetness: No | 0
  Day 28: Portability: number analyzed (Participants) | 13
  Day 28: Portability: Yes | 13
  Day 28: Portability: No | 0

31. Secondary Outcome: Patient Satisfaction During Wear - Interference With Daily Living: Chronic and Dehisced Surgical Wounds Only
Description: Patient satisfaction during wear in interference with daily living at Day 14 and Day 28 measured by response of 'Yes' or 'No' to the following:
  * Showering
  * Sleeping
  * Socializing
  * Working
Time Frame: Day 14 and Day 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 15
Participants
  Day 14: Showering: number analyzed (Participants) | 14
  Day 14: Showering: Yes | 8
  Day 14: Showering: No | 6
  Day 14: Sleeping: Yes | 15
  Day 14: Sleeping: No | 0
  Day 14: Socializing: Yes | 14
  Day 14: Socializing: No | 1
  Day 14: Working: number analyzed (Participants) | 14
  Day 14: Working: Yes | 7
  Day 14: Working: No | 7
  Day 28: Showering: number analyzed (Participants) | 13
  Day 28: Showering: Yes | 8
  Day 28: Showering: No | 5
  Day 28: Sleeping: number analyzed (Participants) | 13
  Day 28: Sleeping: Yes | 13
  Day 28: Sleeping: No | 0
  Day 28: Socializing: number analyzed (Participants) | 13
  Day 28: Socializing: Yes | 12
  Day 28: Socializing: No | 1
  Day 28: Working: number analyzed (Participants) | 13
  Day 28: Working: Yes | 8
  Day 28: Working: No | 5

32. Secondary Outcome: Ease of Application and Removal: Chronic and Dehisced Surgical Wounds Only
Description: Ease of application and removal of the PICO 14 dressing for Chronic and Dehisced Surgical Wounds determined by overall count of dressings applied/removed based on responses to the questions "Was it easy to apply the dressing" and "Was it easy to remove the dressing" as either 'Yes' or 'No'.
Time Frame: Up to 28 days
Population: as for outcome 16
Measure: Count of Units; unit: dressings
Units Other Than Participants: dressings
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Number analyzed (dressings) | 113
dressings
  Was it easy to apply the dressing: Yes | 112
  Was it easy to apply the dressing: No | 1
  Was it easy to remove the dressing: number analyzed (dressings) | 109
  Was it easy to remove the dressing: Yes | 105
  Was it easy to remove the dressing: No | 4

33. Secondary Outcome: Dressing Wear Time: Chronic and Dehisced Surgical Wounds Only
Description: Dressing wear time in days summarized for Chronic and Dehisced Surgical Wounds over the treatment period up to 28 days.
Time Frame: Up to 28 days
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: dressings
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Number analyzed (dressings) | 114
days | 3.6 (2.0)

34. Secondary Outcome: Dressing Conformability: Chronic and Dehisced Surgical Wounds Only
Description: Dressing conformability to the wound measured by the number of responses to the question "Was the dressing conformable on the incision/wound?" as either 'Yes' or 'No'.
Time Frame: Up to 28 days
Population: as for outcome 16
Measure: Count of Units; unit: dressings
Units Other Than Participants: dressings
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Number analyzed (dressings) | 112
dressings
  Yes | 112
  No | 0

35. Secondary Outcome: Number of Dressings Used: Chronic and Dehisced Surgical Wounds Only
Description: Dressing change frequency summarized as the number of dressings used per participant for Chronic and Dehisced Surgical Wounds
Time Frame: Up to 28 days
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: dressings per participant
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
dressings per participant | 7.1 (3.3)

36. Secondary Outcome: Reason for Dressing Change: Chronic and Dehisced Surgical Wounds Only
Description: Reason for dressing change for Chronic and Dehisced Surgical Wounds only. Count of occurrences by dressing were categorized as 'Yes' or 'No':
  * Routine dressing change
  * Inadequate exudate management
  * Pain/discomfort
  * Dressing damaged
  * Dressing fell off
  * Patient removed dressing
  * Adverse Event
  * Surgical procedure
  * Safety alarm
  * Dressing components not in place
  * No vacuum
  * other
Time Frame: Up to 28 days
Population: as for outcome 16
Measure: Count of Units; unit: dressings
Units Other Than Participants: dressings
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 16
Number analyzed (dressings) | 114
dressings
  Routine dressing change: Yes | 84
  Routine dressing change: No | 30
  Inadequate exudate management: Yes | 8
  Inadequate exudate management: No | 106
  Pain/discomfort: Yes | 0
  Pain/discomfort: No | 114
  Dressing damaged: Yes | 0
  Dressing damaged: No | 114
  Dressing fell off: Yes | 3
  Dressing fell off: No | 111
  Patient removed dressing: Yes | 0
  Patient removed dressing: No | 114
  Adverse Event: Yes | 2
  Adverse Event: No | 112
  Surgical procedure: Yes | 0
  Surgical procedure: No | 114
  Safety alarm: Yes | 2
  Safety alarm: No | 112
  Dressing components not in place: Yes | 0
  Dressing components not in place: No | 114
  No vacuum: Yes | 3
  No vacuum: No | 111
  Other: Yes | 17
  Other: No | 97

37. Secondary Outcome: Clinician Acceptability of PICO 14 at Discontinuation of Therapy: Chronic and Dehisced Surgical Wounds Only
Description: Acceptability of the device determined from the clinician's response (Yes/No) at discontinuation of therapy by participant (i.e., Day 28) to the question: Overall are you satisfied with the performance of the PICO 14 system (pump and PICO 14 dressing)?
Time Frame: Day 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | PICO 14 Chronic/Dehisced Surgical Wounds
Number analyzed (Participants) | 13
Participants
  Yes | 13
  No | 0

ADVERSE EVENTS:
Time Frame: Adverse events for closed incisions collected 14 days post-surgery with a further 16 days follow-up period, up to 30 days from initial application of treatment. Adverse events for chronic wounds and dehisced surgical wounds were collected up to 28 days during the therapy period with no follow up.
Arm/Group | PICO 14 Closed Incisions | PICO 14 Chronic/Dehisced Surgical Wounds
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/19
Serious Adverse Events (participants affected / at risk) | 1/25 | 3/19
Other Adverse Events (participants affected / at risk) | 21/25 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PICO 14 Closed Incisions (N=25) | PICO 14 Chronic/Dehisced Surgical Wounds (N=19)
ANEMIA (Blood and lymphatic system disorders) | 1 | 0
ADMITTED TO HOSPITAL WITH A CHEST INFECTION. (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PATIENTS GENERAL HEALTH HAS QUICKLY DECLINED AND IS NOW AT END OF LIFE (General disorders) | 0 | 1
PATIENT HOSPITALISED WITH CHEST PAIN (General disorders) | 0 | 1
WOUND INFECTION (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PICO 14 Closed Incisions (N=25) | PICO 14 Chronic/Dehisced Surgical Wounds (N=19)
ABDOMINAL DISCOMFORT (General disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0
ANAEMIA POST SURGERY (Blood and lymphatic system disorders) | 1 | 0
BLISTER ON RIGHT EDGE OF ADHESIVE STRIP (Skin and subcutaneous tissue disorders) | 1 | 0
BLISTER TO BELLY BUTTON (Skin and subcutaneous tissue disorders) | 1 | 0
BLOOD STAINED SPUTUM (Vascular disorders) | 1 | 0
BP 106/47- HYPOTENSION (General disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0
CHEST INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CONGESTIVE DERMATITIS OF THE LOWER LEGS (Skin and subcutaneous tissue disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
DISTENDED ABDOMEN (Gastrointestinal disorders) | 1 | 0
DRAIN SITE OOZING PUS AND RED (General disorders) | 1 | 0
DRESSING STUCK TO THE WOUND AND CAUSED SOME EXCORIATION TO THE SURROUNDING SKIN (Skin and subcutaneous tissue disorders) | 0 | 1
DROWSINESS (Nervous system disorders) | 1 | 0
ELEVATED INFLAMMATORY MARKERS (General disorders) | 1 | 0
ELEVATED WHITE BLOOD CELL COUNT POST-OPERATIVELY (Blood and lymphatic system disorders) | 1 | 0
EXCORIATION TO SURROUNDING SKIN TO WOUND (Skin and subcutaneous tissue disorders) | 0 | 1
EXTENSIVE BRUISING TO OPERATED LEG (Vascular disorders) | 1 | 0
FAINT DAY 9 POST-OPERATIVELY (Nervous system disorders) | 1 | 0
FALL AT HOME- HIT HEAD (Injury, poisoning and procedural complications) | 1 | 0
FEELING GENERALLY UNWELL (Psychiatric disorders) | 1 | 0
FEELING ROUGH (General disorders) | 1 | 0
FRANK RECTAL BLEED (Gastrointestinal disorders) | 1 | 0
HAEMATOMA AT WOUND SITE (Vascular disorders) | 1 | 0
HAEMATURIA ON CATHETER REMOVAL (Renal and urinary disorders) | 1 | 0
HB 97 (Blood and lymphatic system disorders) | 1 | 0
HEADACHES (Nervous system disorders) | 1 | 0
HYPERGLYCAEMIA (Endocrine disorders) | 1 | 0
HYPOGLYCEMIA (Endocrine disorders) | 1 | 0
HYPOKALAEMIA (Endocrine disorders) | 1 | 0
HYPOTENSION (General disorders) | 1 | 0
ILEOSTOMY LEAK INTO WOUND DRESSING (Gastrointestinal disorders) | 1 | 0
ILEUS (General disorders) | 3 | 0
INFECTED HAEMATOMA (Vascular disorders) | 1 | 0
LEFT ELBOW PAIN. NUMBNESS TI RING & LITTLE FINGER (General disorders) | 1 | 0
LOOSE BOWELS (Gastrointestinal disorders) | 1 | 0
LOOSE STOOL (Gastrointestinal disorders) | 1 | 0
LOOSE STOOL INCONTINENCE (Gastrointestinal disorders) | 0 | 1
LOW EGFR (Renal and urinary disorders) | 1 | 0
LOW MAGNESIUM (Endocrine disorders) | 2 | 0
LOW PHOSPHATE (Endocrine disorders) | 1 | 0
LOW POST-OPERATIVE SODIUM (Blood and lymphatic system disorders) | 2 | 0
LOW POTASSIUM (Endocrine disorders) | 1 | 0
LOW SODIUM LEVEL (Endocrine disorders) | 1 | 0
LOW TEMPERATURE (General disorders) | 1 | 0
MACERATED WOUND EDGES (Skin and subcutaneous tissue disorders) | 0 | 1
MELENA (Gastrointestinal disorders) | 1 | 0
MIGRAINE (Nervous system disorders) | 1 | 0
MILD CRAMPS (Musculoskeletal and connective tissue disorders) | 1 | 0
MILD PAIN (General disorders) | 2 | 0
MONOCYTES: 0.9 HB: 102 WBC: 14.7 NEUTROPHILS: 11.7 CREATINE: 91 E-GFR/1.73M*2 50 (Immune system disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 11 | 0
NONE PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OEDEMA- ANKLES (General disorders) | 1 | 0
ON ARRIVAL WAS FOUND TO HAVE 2 X MOISTURE LESIONS TO SKIN (Skin and subcutaneous tissue disorders) | 0 | 1
OOZING DRAIN WOUND SITE (General disorders) | 1 | 0
PAIN (Gastrointestinal disorders) | 3 | 0
PAIN AROUND WOUND SITE AFTER REMOVAL OF CLIPS (General disorders) | 1 | 0
PAIN CENTRAL ABDOMEN (Gastrointestinal disorders) | 1 | 0
PAIN ON REMOVAL OF DRESSING (General disorders) | 0 | 1
PAIN OPERATED SITE (Injury, poisoning and procedural complications) | 1 | 0
PAIN OPERATIVE SITE (General disorders) | 1 | 0
PAIN RIGHT SIDE (General disorders) | 1 | 0
PAIN VAS 6-8 IN OPERATED KNEE (General disorders) | 1 | 0
PAINFUL FOOT WHEN TWISTED ANKLE DURING A FALL (Injury, poisoning and procedural complications) | 0 | 1
PANIC ATTACKS (Psychiatric disorders) | 1 | 0
PARTICIPANT FINDING PICO14 DRESSING UNCOMFOTABLE, DISTURBING SLEEP (General disorders) | 0 | 1
PAIN FROM COCCYX NOT WOUND SITE AS ADHESIVE STRIPS TOUCH COCCYX (PAIN IN COCCYX FROM PREVIOUS FALL) (General disorders) | 0 | 1
PASSED FRESH BLOOD PER RECTUM (Gastrointestinal disorders) | 1 | 0
PATIENT DESCRIBES INTERMITTENT COOLING SENSATION ON FOOT OF OPERATED LEG (Nervous system disorders) | 1 | 0
PATIENT HAD COVID (Infections and infestations) | 0 | 1
PATIENT PRESENTED AND TREATED FOR ONGOING EXACERBATED COPD SYMPTOMS & SUSPECTED CHEST INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
POOR URINE OUTPUT (Renal and urinary disorders) | 1 | 0
POST-OPERATIVE ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
POST-OPERATIVE ITCH (Skin and subcutaneous tissue disorders) | 1 | 0
POSTURAL DROP HYPOTENSION (General disorders) | 1 | 0
PRESSURE DAMAGE TO THE DORSAL CREASE FROM STOCKING MOVEMENT AND CREASING OVER AREA (Injury, poisoning and procedural complications) | 0 | 1
RAISED BLOOD SUGAR 9.6 (Endocrine disorders) | 1 | 0
RAISED C-REACTIVE PROTEIN (General disorders) | 1 | 0
RAISED CREATININE (Renal and urinary disorders) | 1 | 0
RAISED POST-OPERATIVE WHITE BLOOD CELLS (General disorders) | 1 | 0
RAISED RED BLOOD COUNT (Blood and lymphatic system disorders) | 1 | 0
RAISED WHITE BLOOD COUNT (Immune system disorders) | 2 | 0
RECTAL BLEED (Gastrointestinal disorders) | 1 | 0
REDDEN AREA LEFT HEEL DUE TO PRESSURE, SKIN IS NOT BROKEN (Skin and subcutaneous tissue disorders) | 1 | 0
REDUCED O2 SATURATIONS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SEVERE ITCHING ON SURGICAL SITE (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN IRRITATION UNDER THE BANDAGE (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN RASH FORMED POST-OP, CLUSTERED IN DENSE LINES & AREAS OF SKIN ACROSS RIGHT-SID CHEST & SHOULDER (Skin and subcutaneous tissue disorders) | 1 | 0
SLIGHT POST-OPERATIVE ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
SLUGGISH BOWEL (Gastrointestinal disorders) | 1 | 0
SMALL BOWEL LOOP OBSTRUCTION (General disorders) | 1 | 0
SMALL BRUISING/DEEP TISSUE INJURY TO LEFT EDGE OF WOUND (Skin and subcutaneous tissue disorders) | 0 | 1
SORE NOSE DUE TO NASOJEJUNAL AND NASOGASTRIC TUBE (General disorders) | 1 | 0
SUPERFICIAL WOUND DEHISCENE (General disorders) | 1 | 0
SWELLING LOWER LEG (General disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 3 | 0
TRAUMA TO WOUND BED ON REMOVAL OF DRESSING (Skin and subcutaneous tissue disorders) | 0 | 1
TYPE 7 STOOL- DIARRHEA (Gastrointestinal disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
URINARY TRACT INFECTION (Renal and urinary disorders) | 2 | 0
URINE CONCENTRATED (Renal and urinary disorders) | 2 | 0
VACANT EPISODE (Nervous system disorders) | 1 | 0
VASOVAGAL (Nervous system disorders) | 1 | 0
VERY DIZZY (Nervous system disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 5 | 0
VOMITTED GREEN FLUID (Gastrointestinal disorders) | 1 | 0
WHITE CELL COUNT ELEVATED POST-OPERATIVELY (Blood and lymphatic system disorders) | 1 | 0
WIND LIKE UPPER ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
WIND PAIN (Gastrointestinal disorders) | 1 | 0
WOUND INFECTION (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT05234632/Prot_SAP_000.pdf